CLINICAL TRIAL: NCT00297102
Title: Effect of Roflumilast on Exacerbation Rate in Patients With COPD. The AURA Study
Brief Title: Effect of Roflumilast on Exacerbation Rate in Patients With Chronic Obstructive Pulmonary Disease (COPD): The AURA Study (BY217/M2-124)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-124
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Roflumilast; COPD; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roflumilast (Active Comparator): 500 mcg, once daily, oral administration in the morning
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 500 mcg, once daily, oral administration in the morning
  Arms: Roflumilast
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the effect of roflumilast on exacerbation rate and pulmonary function in patients with chronic obstructive pulmonary disease (COPD). Roflumilast will be administered orally once daily in the morning at one dose level. The study duration will last up to 56 weeks. The study will provide further data on safety and tolerability of roflumilast.

For additional information (for US patients only) see www.COPDSTUDY.net or dial 866-788-2673 (toll free).

ELIGIBILITY:
Main Inclusion Criteria:

* COPD patients having at least one exacerbation within last year
* FEV1/FVC ratio (post-bronchodilator) ≤ 70%
* FEV1 (post-bronchodilator) ≤ 50% of predicted

Main Exclusion Criteria:

* COPD exacerbation not resolved at first baseline visit
* Diagnosis of asthma and/or other relevant lung disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1523 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (149):
- United States (46):
  - Altana Pharma/Nycomed Investigational Site, Fullerton, California
  - Altana Pharma/Nycomed Investigational Site, Los Angeles, California
  - Altana Pharma/Nycomed Investigational Site, Palmdale, California
  - Altana Pharma/Nycomed Investigational Site, Rancho Mirage, California
  - Altana Pharma/Nycomed Investigational Site, San Diego, California
  - Altana Pharma/Nycomed Investigational Site, Bay Pines, Florida
  - Altana Pharma/Nycomed Investigational Site, Miami, Florida
  - Altana Pharma/Nycomed Investigational Site, Panama City, Florida
  - Altana Pharma/Nycomed Investigational Site, Atlanta, Georgia
  - Altana Pharma/Nycomed Investigational Site, Marietta, Georgia
  - Altana Pharma/Nycomed Investigational Site, Hines, Illinois
  - Altana Pharma/Nycomed Investigational Site, South Bend, Indiana
  - Altana Pharma/Nycomed Investigational Site, Lebanon, Kentucky
  - Altana Pharma/Nycomed Investigational Site, Metairie, Louisiana
  - Altana Pharma/Nycomed Investigational Site, New Orleans, Louisiana
  - Altana Pharma/Nycomed Investigational Site, Slidell, Louisiana
  - Altana Pharma/Nycomed Investigational Site, Sunset, Louisiana
  - Altana Pharma/Nycomed Investigational Site, Bangor, Maine
  - Altana Pharma/Nycomed Investigational Site, Baltimore, Maryland
  - Altana Pharma/Nycomed Investigational Site, North Dartmouth, Massachusetts
  - Altana Pharma/Nycomed Investigational Site, Edina, Minnesota
  - Altana Pharma/Nycomed Investigational Site, Minneapolis, Minnesota
  - Altana Pharma/Nycomed Investigational Site, Chesterfield, Missouri
  - Altana Pharma/Nycomed Investigational Site, St Louis, Missouri
  - Altana Pharma/Nycomed Investigational Site, Billings, Montana
  - Altana Pharma/Nycomed Investigational Site, Missoula, Montana
  - Altana Pharma/Nycomed Investigational Site, Lincoln, Nebraska
  - Altana Pharma/Nycomed Investigational Site, Omaha, Nebraska
  - Altana Pharma/Nycomed Investigational Site, Reno, Nevada
  - Altana Pharma/Nycomed Investigational Site, Cherry Hill, New Jersey
  - Altana Pharma/Nycomed Investigational Site, Springfield, New Jersey
  - Altana Pharma/Nycomed Investigational Site, New York, New York
  - Altana Pharma/Nycomed Investigational Site, Winston-Salem, North Carolina
  - Altana Pharma/Nycomed Investigational Site, Cincinnati, Ohio
  - Altana Pharma/Nycomed Investigational Site, Columbus, Ohio
  - Altana Pharma/Nycomed Investigational Site, Toledo, Ohio
  - Altana Pharma/Nycomed Investigational Site, Youngstown, Ohio
  - Altana Pharma/Nycomed Investigational Site, Lake Oswego, Oregon
  - Altana Pharma/Nycomed Investigational Site, Philadelphia, Pennsylvania
  - Altana Pharma/Nycomed Investigational Site, Cranston, Rhode Island
  - Altana Pharma/Nycomed Investigational Site, East Providence, Rhode Island
  - Altana Pharma/Nycomed Investigational Site, Austin, Texas
  - Altana Pharma/Nycomed Investigational Site, Dallas, Texas
  - Altana Pharma/Nycomed Investigational Site, Charlottesville, VA, Virginia
  - Altana Pharma/Nycomed Investigational Site, Bellingham, Washington
  - Altana Pharma/Nycomed Investigational Site, Marietta, Wisconsin
- Australia (11):
  - Altana Pharma/Nycomed Investigational Site, Adelaide South Australia
  - Altana Pharma/Nycomed Investigational Site, Box Hill
  - Altana Pharma/Nycomed Investigational Site, Camperdown
  - Altana Pharma/Nycomed Investigational Site, Clayton
  - Altana Pharma/Nycomed Investigational Site, Concord
  - Altana Pharma/Nycomed Investigational Site, Geelong
  - Altana Pharma/Nycomed Investigational Site, Kippa-Ring
  - Altana Pharma/Nycomed Investigational Site, Nedlands
  - Altana Pharma/Nycomed Investigational Site, South Brisbane
  - Altana Pharma/Nycomed Investigational Site, Toorak Gardens
  - Altana Pharma/Nycomed Investigational Site, Wayville
- Austria (7):
  - Altana Pharma/Nycomed Investigational Site, Feldbach
  - Altana Pharma/Nycomed Investigational Site, Gänserndorf
  - Altana Pharma/Nycomed Investigational Site, Hallein
  - Altana Pharma/Nycomed Investigational Site, Innsbruck
  - Altana Pharma/Nycomed Investigational Site, Linz
  - Altana Pharma/Nycomed Investigational Site, Natters
  - Altana Pharma/Nycomed Investigational Site, Spittal an der Drau
- Brazil (12):
  - Altana Pharma/Nycomed Investigational Site, Belo Horizonte - MG CEP
  - Altana Pharma/Nycomed Investigational Site, Botucatu - SP CEP
  - Altana Pharma/Nycomed Investigational Site, Curitiba-PR
  - Altana Pharma/Nycomed Investigational Site, Florianópolis-SC
  - Altana Pharma/Nycomed Investigational Site, Juiz de Fora-MG
  - Altana Pharma/Nycomed Investigational Site, Porto Alegre
  - Altana Pharma/Nycomed Investigational Site, Porto Alegre-RS
  - Altana Pharma/Nycomed Investigational Site, Quadra 605 Brasilia - DF
  - Altana Pharma/Nycomed Investigational Site, Recife - PE
  - Altana Pharma/Nycomed Investigational Site, Rio de Janeiro-RJ
  - Altana Pharma/Nycomed Investigational Site, Santo André-SP
  - Altana Pharma/Nycomed Investigational Site, São Paulo-SP
- France (25):
  - Altana Pharma/Nycomed Investigational Site, Beuvry
  - Altana Pharma/Nycomed Investigational Site, Chauny
  - Altana Pharma/Nycomed Investigational Site, Clermont-Ferrand Cedex1
  - Altana Pharma/Nycomed Investigational Site, Ferolles-Attily
  - Altana Pharma/Nycomed Investigational Site, Grasse
  - Altana Pharma/Nycomed Investigational Site, La Teste-de-Buch
  - Altana Pharma/Nycomed Investigational Site, Lens
  - Altana Pharma/Nycomed Investigational Site, Libourne
  - Altana Pharma/Nycomed Investigational Site, Lille
  - Altana Pharma/Nycomed Investigational Site, Lyon
  - Altana Pharma/Nycomed Investigational Site, Marcq-en-Barœul
  - Altana Pharma/Nycomed Investigational Site, Martigues
  - Altana Pharma/Nycomed Investigational Site, Metz
  - Altana Pharma/Nycomed Investigational Site, Montigny-lès-Metz
  - Altana Pharma/Nycomed Investigational Site, Montpellier
  - Altana Pharma/Nycomed Investigational Site, Nice
  - Altana Pharma/Nycomed Investigational Site, Nîmes
  - Altana Pharma/Nycomed Investigational Site, Ollioules
  - Altana Pharma/Nycomed Investigational Site, Paris
  - Altana Pharma/Nycomed Investigational Site, Perpignan
  - Altana Pharma/Nycomed Investigational Site, Saint-Etienne
  - Altana Pharma/Nycomed Investigational Site, Saint-Laurent-du-Var
  - Altana Pharma/Nycomed Investigational Site, Saint-Quentin
  - Altana Pharma/Nycomed Investigational Site, Toulon
  - Altana Pharma/Nycomed Investigational Site, Vieux-Condé
- Germany (6):
  - Altana Pharma/Nycomed Investigational Site, Deggendorf
  - Altana Pharma/Nycomed Investigational Site, Fulda
  - Altana Pharma/Nycomed Investigational Site, Kassel
  - Altana Pharma/Nycomed Investigational Site, Lübeck
  - Altana Pharma/Nycomed Investigational Site, Marburg
  - Altana Pharma/Nycomed Investigational Site, Schwetzingen
- Hungary (11):
  - Altana Pharma/Nycomed Investigational Site, Balassagyarmat
  - Altana Pharma/Nycomed Investigational Site, Budapest
  - Altana Pharma/Nycomed Investigational Site, Debrecen
  - Altana Pharma/Nycomed Investigational Site, Gyula
  - Altana Pharma/Nycomed Investigational Site, Komárom
  - Altana Pharma/Nycomed Investigational Site, Mosdós
  - Altana Pharma/Nycomed Investigational Site, Mosonmagyaróvár
  - Altana Pharma/Nycomed Investigational Site, Nyiregyháza
  - Altana Pharma/Nycomed Investigational Site, Pécs
  - Altana Pharma/Nycomed Investigational Site, Szeged
  - Altana Pharma/Nycomed Investigational Site, Tapolca
- Altana Pharma/Nycomed Investigational Site, Tauranga, New Zealand
- Altana Pharma/Nycomed Investigational Site, Bucharest, Romania
- Russia (2):
  - Altana Pharma/Nycomed Investigational Site, Moscow
  - Altana Pharma/Nycomed Investigational Site, Saint Petersburg
- United Kingdom (27):
  - Altana Pharma/Nycomed Investigational Site, Baillieston, Glasgow
  - Altana Pharma/Nycomed Investigational Site, Bangor, Northern Ireland
  - Altana Pharma/Nycomed Investigational Site, Bath
  - Altana Pharma/Nycomed Investigational Site, Bath, Avon
  - Altana Pharma/Nycomed Investigational Site, Belfast
  - Altana Pharma/Nycomed Investigational Site, Birmingham
  - Altana Pharma/Nycomed Investigational Site, Chesterfield
  - Altana Pharma/Nycomed Investigational Site, Co. Antrim
  - Altana Pharma/Nycomed Investigational Site, Cottingham, E York
  - Altana Pharma/Nycomed Investigational Site, County Antrim
  - Altana Pharma/Nycomed Investigational Site, Downpatrick, Northern Ireland
  - Altana Pharma/Nycomed Investigational Site, East Sussex
  - Altana Pharma/Nycomed Investigational Site, Fife
  - Altana Pharma/Nycomed Investigational Site, Glasgow
  - Altana Pharma/Nycomed Investigational Site, Glengormley Newtownabbey
  - Altana Pharma/Nycomed Investigational Site, Harrow
  - Altana Pharma/Nycomed Investigational Site, Kent
  - Altana Pharma/Nycomed Investigational Site, Liverpool
  - Altana Pharma/Nycomed Investigational Site, Nottingham
  - Altana Pharma/Nycomed Investigational Site, Randalstown
  - Altana Pharma/Nycomed Investigational Site, Royal Leamington Spa
  - Altana Pharma/Nycomed Investigational Site, Sheffield
  - Altana Pharma/Nycomed Investigational Site, Solihull
  - Altana Pharma/Nycomed Investigational Site, Southampton
  - Altana Pharma/Nycomed Investigational Site, Southdown, Bath
  - Altana Pharma/Nycomed Investigational Site, Sunbury on Thames, Middlesex
  - Altana Pharma/Nycomed Investigational Site, Vale of Glamorgan

REFERENCES:
- [Result] Calverley PM, Rabe KF, Goehring UM, Kristiansen S, Fabbri LM, Martinez FJ; M2-124 and M2-125 study groups. Roflumilast in symptomatic chronic obstructive pulmonary disease: two randomised clinical trials. Lancet. 2009 Aug 29;374(9691):685-94. doi: 10.1016/S0140-6736(09)61255-1. PMID 19716960
- [Derived] Facius A, Krause A, Claret L, Bruno R, Lahu G. Modeling and Simulation of Pivotal Clinical Trials Using Linked Models for Multiple Endpoints in Chronic Obstructive Pulmonary Disease With Roflumilast. J Clin Pharmacol. 2017 Aug;57(8):1042-1052. doi: 10.1002/jcph.885. Epub 2017 Apr 17. PMID 28419462
- [Derived] Hanania NA, Calverley PM, Dransfield MT, Karpel JP, Brose M, Zhu H, Goehring UM, Rowe P. Pooled subpopulation analyses of the effects of roflumilast on exacerbations and lung function in COPD. Respir Med. 2014 Feb;108(2):366-75. doi: 10.1016/j.rmed.2013.09.018. Epub 2013 Sep 30. PMID 24120253
- [Derived] Wedzicha JA, Rabe KF, Martinez FJ, Bredenbroker D, Brose M, Goehring UM, Calverley PMA. Efficacy of roflumilast in the COPD frequent exacerbator phenotype. Chest. 2013 May;143(5):1302-1311. doi: 10.1378/chest.12-1489. PMID 23117188
- [Derived] Cazzola M, Picciolo S, Matera MG. Roflumilast in chronic obstructive pulmonary disease: evidence from large trials. Expert Opin Pharmacother. 2010 Feb;11(3):441-9. doi: 10.1517/14656560903555201. PMID 20102307

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Roflumilast | Placebo
Started | 765 (Includes all randomized patients who took at least one dose of the investigational drug.) | 758 (Includes all randomized patients who took at least one dose of the investigational drug.)
Completed | 502 | 525
Not Completed | 263 | 233

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast | Placebo | Total
Number analyzed (Participants) | 765 | 758 | 1523
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.53 (9.5) | 63.36 (9.2) | 63.45 (9.4)
Gender [Count of Participants; unit: Participants]
  Female | 225 | 220 | 445
  Male | 540 | 538 | 1078

OUTCOME MEASURES:

1. Primary Outcome: Pre-bronchodilator Forced Expiratory Volume in First Second (FEV1)
Description: Mean change from baseline during the treatment period in pre-bronchodilator FEV1 [L]
Time Frame: Change from baseline over 52 weeks of treatment
Population: ITT (Intention to Treat) analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 745 | 745
mL | 46 (8) | 8 (8)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; Repeated measurements analysis (change from baseline over 52 weeks of treatment taking all post-randomization measurements into account); Mean Difference (Net) = 39, 95% CI 2-sided [18 to 60], Standard Error of Mean 11

2. Primary Outcome: COPD Exacerbation Rate (Moderate or Severe)
Description: Mean rate of COPD exacerbations requiring oral or parenteral glucocorticosteroids (=moderate COPD exacerbations), or requiring hospitalization, or leading to death (=severe COPD exacerbations), per patient per year. A COPD exacerbation is an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough and/or sputum beyond day-to-day variability sufficient to warrant a change in management [American Thoracic Society (ATS) / European Respiratory Society (ERS) 2005].
Time Frame: 52 weeks treatment period
Population: ITT analysis.
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient per year
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 765 | 758
exacerbations per patient per year | 1.077 [0.960 to 1.207] | 1.266 [1.141 to 1.404]
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.0278, Poisson regression — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; Rate ratio = 0.851, 95% CI 2-sided [0.737 to 0.982], Standard Error of Mean 0.062

3. Secondary Outcome: Post-bronchodilator FEV1 [L]
Description: Mean change from baseline during the treatment period in post-bronchodilator FEV1 [L]
Time Frame: Change from baseline over 52 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 729 | 736
mL | 57 (9) | 8 (8)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 49, 95% CI 2-sided [26 to 71], Standard Error of Mean 11

4. Secondary Outcome: Time to Mortality Due to Any Reason
Time Frame: 52 weeks treatment period
Population: ITT analysis. Number of participants analyzed = number of participants who died.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 17 | 17
days | 213.8 (118.9) | 207.5 (108.5)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.9212, Cox proportional hazards regression — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; Hazard Ratio (HR) = 1.035, 95% CI 2-sided [0.526 to 2.034], Standard Error of Mean 0.357 — The statistical analysis is based on the ITT Analysis Set (n= 765 in the roflumilast group, n= 758 in the placebo group)

5. Secondary Outcome: Natural Log-transformed C-reactive Protein (CRP)
Description: Mean change from baseline to the last post randomization measurement in natural log-transformed CRP
Time Frame: Change from baseline to last post randomization measurement (52 weeks)
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 691 | 694
mg/L | 1.0475 [0.9584 to 1.1450] | 1.1003 [1.0071 to 1.2021]
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.4089, ANCOVA — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; ANCOVA model including last observation carried forward (LOCF) method; Mean Difference calculated as ratio = 0.9521, 95% CI 2-sided [0.8472 to 1.0699]

6. Secondary Outcome: Mean Transition Dyspnea Index (TDI) Focal Score During the Treatment Period
Description: The TDI is a recognized questionnaire to measure dyspnea in an out patient COPD population. At baseline, 3 components of dyspnea, each graded with 4 questions, were asked: - Functional Impairment - Magnitude of Task - Magnitude of Effort At each of the post-randomization visits questions from the TDI were asked related to 3 components: Change in - Functional Impairment - Magnitude of Task - Magnitude of Effort Each question in the TDI is graded from -3 (major deterioration) to +3 (major improvement). This results in a TDI Focal Score ranging from -9 to +9.
Time Frame: Change from baseline over 52 weeks of treatment
Population: ITT analysis. Number of participants analyzed = number of participants with data available.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roflumilast | Placebo
Number analyzed (Participants) | 741 | 745
scores on a scale | 0.658 (0.084) | 0.426 (0.082)
Statistical Analysis 1: Comparison: Roflumilast vs Placebo; Test type: Superiority or Other; p = 0.0356, ANCOVA — No adjustment of the significance level was done as a hierarchical approach for hypotheses testing was used; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.233, 95% CI 2-sided [0.016 to 0.449], Standard Error of Mean 0.111

ADVERSE EVENTS:
Time Frame: 52 weeks treatment period
Description: The Safety Set was based on all randomized patients who took at least one dose of the investigational drug after randomization. 4 patients randomized to placebo received roflumilast instead and were included in the roflumilast group for safety analyses. 1 patient was randomized twice. The second randomization is only included in the Safety Set.
Arm/Group | Roflumilast | Placebo
Serious Adverse Events (participants affected / at risk) | 144/769 | 153/755
Other Adverse Events (participants affected / at risk) | 232/769 | 136/755
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=769) | Placebo (N=755)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 70 (95) | 82 (108)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 7 (7) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 4 (4)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8) | 11 (13)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 2 (4)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (2)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Arterial restenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscoloskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Blepharochalasis (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Bronchoscopy (Investigations) | 0 (0) | 1 (1)
Computerised tomogram thorax abnormal (Investigations) | 0 (0) | 1 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Physical assault (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=769) | Placebo (N=755)
Nasopharyngitis (Infections and infestations) | 57 (76) | 50 (65)
Bronchitis (Infections and infestations) | 33 (41) | 39 (49) — non-serious
Diarrhoea (Gastrointestinal disorders) | 62 (72) | 26 (30) — non-serious
Nausea (Gastrointestinal disorders) | 40 (44) | 15 (15) — non-serious
Weight decreased (Investigations) | 92 (94) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study results may be published and/or presented at scientific meetings. Prior to any submission, all manuscripts/abstracts must be presented to the sponsor for possible comments.